CLINICAL TRIAL: NCT04253730
Title: Characterization of Corticospinal Excitability During Progressive Skin Cooling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr.Gordon Giesbrecht, Professor, University of Manitoba
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E2018:047 (HS21827)
Record Dates: First submitted 2019-11-26; First posted 2020-02-05 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Hypothermia Due to Cold Environment
Keywords: Body Temperature, Skin Temperature, Cooling
MeSH Terms: interventions — Cold-Shock Response

STUDY DESIGN:
Intervention Model Description: Repeat Measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (No Intervention): Subjects will sit at rest wearing a liquid perfused suit containing thermoneutral water for 60 min. The suit will not be turned on during this period.
- Cold Condition (Experimental): Subjects will be cooled for 60-90 min at ~ 4-10°C using a liquid perfused suit. Subjects will then be rewarmed for 30 min at ~ 41°C using the liquid perfused suit.
  Interventions: Other: Cold Stress

INTERVENTIONS:
Other: Cold Stress — 60-90 mins of cooling via a liquid perfused suit circulating ~4-10°C liquid.
  Arms: Cold Condition

SUMMARY:
This study characterizes the changes in corticospinal excitability that accompany basic cold stress via skin cooling that result in reduced skin or core temperature and shivering.

DETAILED DESCRIPTION:
Cold stress is known to impair both fine and gross motor movement. Reductions in performance may have life threatening consequences in survival situations where maintenance of muscle control is necessary. Much of the effects cooling has on muscle performance is directly due to its effects on muscle tissue itself, whereas less is known about the effects on the central nervous system. Therefore, the purpose of the study was to characterize corticospinal excitability that accompanies basic cold stress via progressive skin cooling, resulting in reductions in skin (Tsk) or core (Tco) temperature and shivering.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Right Handed
* Pass Magnetic Stimulation Safety Checklist
* Pass Medical Screening Questionnaire

Exclusion Criteria:

* Left Handed
* Any adverse responses to cold exposure (Raynaud's Syndrome)
* Cardiorespiratory Disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Corticospinal Excitability | at 0, 20, 40, 60 and 90 minutes
  Motor Evoked Potentials (MEP) as a percentage of the maximal compound muscle action potential (Mmax) measured via MEG at the Biceps Brachii will serve as the indices of Corticospinal excitbaility

SECONDARY OUTCOMES:
Change in Spinal Excitability | at 0, 20, 40, 60 and 90 minutes
  Cervicomedullary Motor Evoked Potentials (CMEP) as a percentage of the maximal compound muscle action potential (Mmax) measured via MEG at the Biceps Brachii will serve as the indices of spinal excitability
Change in Skin Temperature | at 0, 20, 40, 60 and 90 minutes
  Mean skin temperature of 7 sites
Change in Core Temperature | at 0, 20, 40, 60 and 90 minutes
  Esophageal temperature is the most accurate method representing the temperature of the heart.
Change in Metabolic Heat Production | at 0, 20, 40, 60 and 90 minutes
  Metabolic heat production serves as an objective way to quantify shivering thermogenesis.

OTHER OUTCOMES:
Change in Peripheral nerve excitability | at 0, 20, 40, 60 and 90 minutes
  Excitability of the peripheral nerve measured via EMG at the biceps brachia ( the maximal compound motor action potential (Mmax).
Change in Maximal Voluntary Contraction of Elbow Flexors | at 0, 20, 40, 60 and 90 minutes
  Maximal Isometric Force of elbow flexors measured in kg of force

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Giesbrecht, PhD, Principal Investigator — University of Manitoba
Locations (1):
- 211 Max Bell Centre, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurrie DMG, Talebian Nia M, Power K, Stecina K, Gardiner P, Lockyer E, Giesbrecht GG. Spinal and corticospinal excitability in response to reductions in skin and core temperatures via whole-body cooling. Appl Physiol Nutr Metab. 2022 Feb;47(2):195-205. doi: 10.1139/apnm-2021-0370. Epub 2021 Sep 28. PMID 34582724